CLINICAL TRIAL: NCT04314830
Title: Unpredictable Perturbations During Gait to Improve Balance Performance, Confidence and Participation in Persons With Hemiparesis at a Chronic Stage: a Pilot Study
Brief Title: Gait Perturbations to Improve Balance Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Responsible Party: Principal Investigator, Cyril Duclos, Associate professor, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CRIR-998-0914
Record Dates: First submitted 2020-03-12; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Hemiparesis;Poststroke/CVA

STUDY DESIGN:
Intervention Model Description: Only the experimental intervention was offered in the second phase of the trial, to the participants who received the control intervention in the first phase
Who Masked: Outcomes Assessor
Masking Description: Outcome measures pretraining were collected pre-randomization. Post-training, the assessors were masked for the arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Gait training without perturbation (Active Comparator): Walking on a treadmill with the same duration as a participants of the experimental arm matched for initial gait speed. Treadmill speed did not change along the training program
  Interventions: Device: Gait training without perturbation
- Gait training with perturbations (Experimental): Walking on a treadmill with perturbations produced by changes in the speed of one of the belt of the split-belt treadmill during one gait cycle. Changes in treadmill speed were applied on the paretic or non-paretic side, with and increase or a decrease of the speed of the belt in various magnitude. Perturbations were either repeated with the same characteristics or with different characteristics. Outside of perturbations, treadmill speed did not change along the training program.
  Interventions: Device: Gait training with perturbations

INTERVENTIONS:
Device: Gait training with perturbations — Changes in speed of one of the belt of the split belt treadmill during swing phase
  Arms: Gait training with perturbations
Device: Gait training without perturbation — Walking on a treadmill with steady belt speed
  Arms: Gait training without perturbation

SUMMARY:
Individuals with stroke have balance and gait deficits. Gait training does improve balance and gait abilities, but adding perturbations may have increase these effects. The objective was to compare the effect gait training with and without perturbations on balance and gait abilities in individuals with hemiparesis due to stroke at a chronic stage.

ELIGIBILITY:
Inclusion Criteria:

* able to walk at a comfortable speed less than 1.0 m/s
* have reduced dynamic balance capacities (as evaluated by the mini-BESTest; score below the 95% confidence interval of the mean score of the corresponding age group of normative data)
* with or without a history of fall
* be able to walk on a treadmill, without external support, such as handrails or walking aid, for at least 1 minute

Exclusion Criteria:

* hemineglect (more than 6 omissions on the bell cancellation test),
* cognitive impairment (Mini-Mental State Examination score under 24/30)
* uncorrected visual deficit or pathologies other than stroke which can affect their gait or balance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Balance capacities | Within the week pre-training
  Score at the mini-Balance Evaluation System Test (mini-BESTest). Score between 0 and 28. Higher scores associated with better balance abilities.
Balance capacities | Within the week post-training
  Score at the mini-Balance Evaluation System Test (mini-BESTest). Score between 0 and 28. Higher scores associated with better balance abilities.
Gait capacities | Within the week pre-training
  Self-selected and fast gait speed measured over 10 meters (10 meter walking test)
Gait capacities | Within the week post-training
  Self-selected and fast gait speed measured over 10 meters (10 meter walking test)

SECONDARY OUTCOMES:
Paretic and non-paretic maximal knee extensor strength | Within the week pre-training
  Measure of isometric, maximal knee extensor strength at each knee, using an instrumented dynamometer (Biodex).
Paretic and non-paretic maximal knee extensor strength | Within the week post-training
  Measure of isometric, maximal knee extensor strength at each knee, using an instrumented dynamometer (Biodex)
Balance confidence | Within the week pre-training
  Score at the Activity-specific Balance Confidence (ABC scale), between 0 and 100%, with 100% indicating better balance confidence
Balance confidence | Within the week post-training
  Score at the Activity-specific Balance Confidence (ABC scale), between 0 and 100%, with 100% indicating better balance confidence
Balance confidence | 6 weeks post training
  Score at the Activity-specific Balance Confidence (ABC scale), between 0 and 100%, with 100% indicating better balance confidence
Community reintegration | Within the week pre-training
  Score at the Reintegration to Normal Living Index (RNLI), between 0 and 22, with 0 indicating total reintegration.
Community reintegration | Within the week post-training
  Score at the Reintegration to Normal Living Index (RNLI), between 0 and 22, with 0 indicating total reintegration.
Community reintegration | 6 weeks post training
  Score at the Reintegration to Normal Living Index (RNLI), between 0 and 22, with 0 indicating total reintegration.

OTHER OUTCOMES:
Satisfaction with gait perturbation intervention | Within the week post-training
  Score at the Short Feedback Questionnaire. Rating from "Not at all" to "Extremely" to 9 questions. No total score. Answers interpreted for each question.
Laboratory gait analysis : kinematics | Within the week pre-training
  Lower-limb joint angles, centre of mass during gait at natural and fast speed and during gait perturbations
Laboratory gait analysis : kinematics | Within the week post-training
  Lower-limb joint angles, centre of mass during gait at natural and fast speed and during gait perturbations
Laboratory gait analysis : kinetics | Within the week pre-training
  Ground reaction forces and centre of pressure during gait at natural and fast speed and during gait perturbations
Laboratory gait analysis : kinetics | Within the week post-training
  Ground reaction forces and centre of pressure during gait at natural and fast speed and during gait perturbations
Laboratory gait analysis : electromyographic activity | Within the week pre-training
  EMG activity of 5 muscle groups (tibialis anterior, soleus, rectus femoris, medial hamstring, paravertebral muscles at L3) bilateraly during gait at natural and fast speed and during gait perturbations
Laboratory gait analysis : electromyographic activity | Within the week post-training
  EMG activity of 5 muscle groups (tibialis anterior, soleus, rectus femoris, medial hamstring, paravertebral muscles at L3) bilateraly during gait at natural and fast speed and during gait perturbations

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Duclos, PhD, Principal Investigator — Université de Montréal - CRIR

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esmaeili V, Juneau A, Dyer JO, Lamontagne A, Kairy D, Bouyer L, Duclos C. Intense and unpredictable perturbations during gait training improve dynamic balance abilities in chronic hemiparetic individuals: a randomized controlled pilot trial. J Neuroeng Rehabil. 2020 Jun 17;17(1):79. doi: 10.1186/s12984-020-00707-0. PMID 32552850